CLINICAL TRIAL: NCT06078826
Title: The Effect of Passive Music Therapy and Foot Massage on Hemodynamic Status, Anxiety and Pain Level Applied to Intensive Care Patients ın Tracheal Aspiration Process
Brief Title: The Effect of Passive Music Therapy and Foot Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Pınar TEKİNSOY KARTIN, Associate professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pinar
Record Dates: First submitted 2023-09-07; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Intensive Care Patients
Keywords: Music therapy; Foot massage; Pain; Anxiety; Intensive care
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The research is planned as a prospective, randomized controlled, single-blind, experimental study. The research will be carried out in the 3rd Level Intensive Care Units of Ömer Halisdemir University Training and Research Hospital located in Niğde City Center. The population of this study will consist of patients receiving mechanical ventilator support, who are intubated in the 3rd Level Intensive Care Units of Ömer Halisdemir University Training and Research Hospital in the city center of Niğde. The sample of the study was 'The Effect of Foot Massage on Pain of the Intensive Care Patients:A Parallel Randomized Single-Blind Controlled' study by Momeni et al. (2020), based on pain, power :0.90, type II- error 10%, confidence When the range of 1.96 is taken as a reference, the experimental groups that should be taken as a minimum were calculated as 25 and the control group 25 as a total of 75 patients.
Who Masked: Participant
Masking Description: Patients who meet the research criteria will be numbered after they are determined by the researcher. It will be determined and recorded by the researcher in the digital randomization environment (https://www.randomizer.org/ internet address), which is a simple randomization method, where the enumerated patients will be assigned to the intervention or control group. After randomization, passive music therapy and foot massage will be applied to the patients in the intervention group, and no treatment will be given to the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- passive music therapy group (Experimental): Intubated patients on mechanical ventilator hospitalized in the 3rd Stage Intensive Care Unit will be included in the intervention group 48 hours after admission. The data of the individuals will be collected by face-to-face interview method in the "Ramsey Sedation Scale", "Patient Identification Form", "Patient Follow-up Form", "Behavioral Pain Scale" to determine the level of pain, and "Facial Anxiety Scale" to determine the level of anxiety at the first interview.
  Before the tracheal aspiration procedure, passive music therapy will be applied for 30 minutes and throughout the aspiration, and during this application, music will be continued for approximately two more minutes (15 seconds of first aspiration, 30 seconds of break, 15 seconds of second aspiration) during both aspirations. Patient Follow-up Form, Behavioral Pain Scale and Face Anxiety Scale will be filled again during and after tracheal aspiration (30 minutes later).
  Interventions: Other: passive music therapy
- foot massage group (Experimental): Intubated patients on mechanical ventilator hospitalized in the 3rd Stage Intensive Care Unit will be included in the intervention group 48 hours after admission. The data of the individuals will be collected by face-to-face interview method in the "Ramsey Sedation Scale", "Patient Identification Form", "Patient Follow-up Form", "Behavioral Pain Scale" to determine the level of pain, and "Facial Anxiety Scale" to determine the level of anxiety at the first interview.
  Foot massage will be applied for 30 minutes before the tracheal aspiration process and throughout the aspiration, and the music will be continued for approximately two more minutes (15 seconds of first aspiration, 30 seconds of break, 15 seconds of second aspiration) during both aspirations. Patient Follow-up Form, Behavioral Pain Scale and Face Anxiety Scale will be filled again during and after tracheal aspiration (30 minutes later).
  Interventions: Other: foot massage
- control group (No Intervention): No intervention will be made to the control group, and the routine care practice of the clinic will be applied. "Ramsey Sedation Scale", "Patient Identification Form", "Patient Follow-up Form", "Behavioral Pain Scale" to determine pain level, "Behavioral Pain Scale" to determine the level of anxiety, at the first interview 48 hours after hospitalization in intubated patients hospitalized in the 3rd Stage Intensive Care Unit. Data will be collected by face-to-face interview method, "Face Anxiety Scale". Hemodynamic parameters will be recorded. Patient Follow-up Form, Behavioral Pain Scale and Face Anxiety Scale will be filled again during and after tracheal aspiration (30 minutes later).

INTERVENTIONS:
Other: passive music therapy — 30 minutes before tracheal aspiration to intubated patients connected to mechanical ventilator treated in the 3rd step intensive care unit. and music between 60-74 dB will be played via headphones and MP3 player during aspiration (Şahin, 2018). This music is a 30-minute Hüseyni makam mp3 music recording . Hüseyni makam is effective in the morning and at dawn, and its effect is high between morning and noon. For this reason, passive music therapy practice in the research will be done by the researcher in the morning and afternoon. This maqam has beauty, benevolence, silence, comfort, a sense of peace and a refreshing feature. It has positive effects on the liver, heart, internal organs and spirit and unites with nature.
  Arms: passive music therapy group
Other: foot massage — Massage will be applied by the researcher in the research. Towel, sponge, etc. under the foot to be worked on. The foot will be held at a 45 degree angle While applying, 1-2 drops of liquid Vaseline will be used to moisten the hand. A total of 30 minutes of foot massage will be made for each individual, 15 minutes per foot. Foot massage will start 30 minutes before the start of aspiration and massage will continue throughout the aspiration period. Since the speed of the massage movements and the number of repetitions should be at the normal frequency, the massage will be done at a speed that does not disturb the individual, has a non-stimulating and calming effect and does not tire the practitioner. In the massage, efflorescence (stroking), petrissage and friction (circular rubbing) movements that support circulation and relax the tissues will be used. Evaluations will be made before the foot massage, at the end of the foot massage and 30 minutes after the foot massage.
  Arms: foot massage group

SUMMARY:
Patients hospitalized in tertiary intensive care units are connected to mechanical ventilators due to multiorgan failure, chronic diseases, respiratory failure, etc. Endotracheal aspiration is then necessary to maintain respiratory patency. However, patients feel a lot of pain during this application. Pharmacological methods for pain relief are mostly used in intensive care units. These methods can have many complications. In this study, it was aimed to determine the effect of passive music therapy and foot massage, which are non-pharmacological methods, on hemodynamic status in relieving pain and anxiety that may develop due to this. Reducing the use of pharmacological methods and switching to non-pharmacological methods in pain relief will increase the quality of patient care and recovery results.

This research will be conducted as a prospective, randomized controlled, single-blind, experimental. In the study, passive music therapy will be applied to one of the intervention groups and foot massage will be applied to the other in the tracheal aspiration process, and no application will be made to the control group. Passive music therapy and foot massage will be applied for 30 minutes during the tracheal aspiration procedure. Evaluation will be made before, during and after the application.

When the literature is examined, there are few studies examining the effect of foot massage in intensive care patients, but no studies evaluating the effect of foot massage during the aspiration procedure have been found. For this reason, it is thought that passive music therapy and foot massage applied in the aspiration process in intensive care patients will reduce the level of pain and anxiety, thus positively affecting the hemodynamic status of the patient, increasing the comfort of the patient and improving the results of nursing care. Thus, it is planned to bring an original study that has not been done on the subject to the literature.

DETAILED DESCRIPTION:
Intensive care units are defined as all the methods used to support the patients, to treat the causes of the disease, and to ensure the survival of the patient until the negative results of the partially or completely lost system and/or organ functions are recovered (Şahinoğlu, 2003). Patients in need of intensive care, who have reached the limit of their lives due to an advanced disease, trauma, poisoning, or surgery due to an advanced disease, trauma, poisoning, or surgery, and who need the help of different supportive biomedical devices, are given continuous and high-quality care, and to provide the best outcomes. They are patients who require the health care team to make sacrifices and efforts (Şahinoğlu, 2003; Hatipoğlu, 2002; Wunsch et al., 2004; Clark and Normile, 2000).

Endotracheal tube and mechanical ventilation are life-saving applications in complicated, conscious and unconscious patients with multi-organ failure, who have lost their physiological balance (Craven et. al., 2009). Tracheotomy or the presence of an endotracheal tube in intensive care patients is the process of giving the air that the patient breathes without being filtered, heated and humidified (Ferreira, 2013). Being immobilized for a long time due to the use of sedation in intensive care patients can also cause loss of ciliary movement and cough reflex function, which are natural defense mechanisms. For these reasons, in patients with endotracheal tube, both the secretion of secretions in the respiratory tract increases and the secretions can accumulate in the respiratory tract, causing mechanical obstructions because the patients cannot discharge their secretions. In order to prevent endotracheal tube obstructions and to maintain airway patency, it is extremely important and necessary to aspirate according to the patient's needs (Guglielminotti et al, 2000; Majett, 2013). However, the frequently used, invasive, life-saving endotracheal aspiration procedure brings many undesirable conditions in intensive care patients. The patient has many symptoms such as discomfort, pain, bleeding, infection, bronchospasm, cardiovascular instability, hypoxia/hypoxemia, tracheal or bronchial mucosal damage, change in cerebral blood flow, increase in intracranial pressure, decrease in dynamic lung compliance and residual capacity, atelectasis, hypotension, hypertension. As it may result in complications, unmanaged pain can also cause anxiety as physiological, psychological and behavioral stressors (Gülsoy, 2017; Çelik et al, 2016). Endotracheal aspiration, which is found to be the most painful intervention experienced by intensive care patients in the literature, causes deterioration of comfort, frightening and unpleasant sensations, namely anxiety. It also creates a feeling of suffocation or is expressed as a loss of breathing (Day et al, 2002; Pedersen et al, 2009; Yaman Aktaş, 2013).

Pain assessment and adequate pain management are extremely important, as pain is a major stressor in intensive care patients (Rotonti et al, 2002). If an effective pain management cannot be achieved, physiological, metabolic and behavioral responses occur due to this pain and pain sensation. Increases in heart rate, respiratory rate and blood pressure occur due to catecholamine, glucagon and steroids released due to painful stimuli. However, with the continuation of the painful stimulus, myocardial oxygen consumption increases, saturation decreases, and arrhythmias are observed (Gelinas, 2010; Dikmen, 2012).

The American Society for Pain Management Nursing (ASPMN) reports that pain management of patients who experience interventional pain should be provided at an optimal level before, during and after the intervention, the level of pain and anxiety should be minimized and appropriate nursing interventions should be applied (Yaman Aktas, 2013). Pharmacological and non-pharmacological methods are applied in the management of patients' pain and comfort for invasive procedures. Pharmacological methods such as local anesthetics, non-opioid analgesics, opioid analgesics and interventional sedation and relaxation techniques, meditation, dreaming, massage, cold application, positioning, game activities and music therapy are used non-pharmacological methods (Eti Aslan et al, 2003; Cignacco et al. al, 2007). Reasons for using non-pharmacological methods in the management of pain; reducing the need for the use of analgesics and increasing the comfort of life by reducing/eliminating the pain of the patient. In addition, nonpharmacological methods; it increases the sense of autonomy by empowering the patient (Özveren, 2011; Yaman Aktaş & Karabulut, 2015). Music therapy and foot massage, which are among the non-pharmacological methods that can be used to relieve pain caused by invasive applications, are simple, valuable and inexpensive adjuvant therapies used in pain control due to their ease of use (Yaman Aktaş and Karabulut, 2015).

Since the language of music is universal, its therapeutic and healing properties have been used throughout history and it continues to be effective today. Music therapy, which is used to maintain and improve mental and physical health, is a simple and natural tool that nurses can apply in pain management due to its ease of use. The use of music therapy increases the patient's ability to endure pain by focusing attention on a stimulus other than pain. In addition, music therapy helps to control pain by removing unpleasant painful stimuli and increasing the secretion of endorphins (Eti Aslan, 2006; Özer et al, 2010; Özveren, 2011).

In the descriptive study of Arroyo-Novoa et al. (2008), in which they investigated the pain levels felt as a result of endotracheal aspiration in patients treated in intensive care, they found that 50% of the patients experienced moderate to severe pain and that pharmacological and/or non-pharmacological methods were effective in relieving patients' pain related to endotracheal aspiration. They concluded that there is a need for further experimental studies. In many studies evaluating the effect of music therapy on pain and anxiety in intensive care patients under mechanical ventilation support, and the reflection of this effect on physiological parameters, it has been concluded that music therapy positively affects both anxiety and pain and the physiological changes caused by pain and anxiety (Güngör Çağlar, 2007). 2018; Şahin, 2018; Uzeli Yılmaz, 2016; Yeşim Yaman 2015; Wong et al, 2021; Amonda Golinda et al., 2021; Isabel et. al., 2016; Ya-Li Huang MM et al., 2021). In the literature, studies on music therapy applied during endotracheal aspiration are limited. Yaman Aktaş (2013) found that the music therapy applied to the patients under mechanical ventilation support during the endotracheal aspiration process controlled the sedation levels of the patients and reduced their pain levels. In the study of Akbaş (2021), after music therapy applied to intensive care patients, there was an increase in GCS values, a decrease in agitation, a decrease in systolic/diastolic blood pressure, pulse, respiratory rate, an increase in oxygen saturation values and tidal volume values in MV. and reported a decrease in the mean values of pain scales.

Massage is expressed as the systematic and generally rhythmic application of hand movements to the soft tissues of the body. The planned and purposeful application of touch improves the relationship between the nurse and the patient, reduces respiratory distress, provides relaxation, and reduces the need for analgesia and sedation. In many studies in the literature examining the effects of massage on various parameters such as pain, edema, nausea, vomiting, fatigue and sleep in cancer, diabetes, dementia and dialysis patients and pregnant women, it has been concluded that foot massage is effective (Özdelikara and Tan, 2014; Korhan et al, 2014; Soyman). , 2009). In the literature, intensive In studies examining the effectiveness of acupressure, back massage, and reflexology alone in reducing the physiological symptoms of anxiety in patients with mechanical ventilation support hospitalized in their units, it was determined that foot massage reduces dyspnea and anxiety and increases the level of comfort in patients (Guven and Karataş 2013; Tiran and Chummun, 2005; Gökçen Gökalp 2018). ). Masoumeh Momeni et al (2021) determined that foot massage has an effect on delirium and consciousness level in intensive care patients. In studies examining foot massage in intensive care patients, it was found that it had a positive effect on hemodynamics such as arterial pressure, heart rate, respiratory rate and oxygen level (Azami et al,2015; Nyayu Nina Putri et al, 2021). Masoumeh Momeni et al. (2020) found that in another study examining the effect of foot massage on pain in intensive care patients, it significantly reduced pain scores. When the literature is examined, there are few studies examining the effect of foot massage in intensive care patients, but no studies evaluating the effect of foot massage during the aspiration procedure have been found.

In line with this information, it is thought that passive music therapy and foot massage applied in the aspiration process in intensive care patients will reduce the level of pain and anxiety, thus positively affecting the hemodynamic status of the patient, increasing the comfort of the patient and improving the results of nursing care.

This study was planned to determine the effects of passive music therapy and foot massage applied during aspiration on patients receiving mechanical ventilation support in the tertiary intensive care unit, on their hemodynamic status, pain and anxiety level.

ELIGIBILITY:
Inclusion Criteria:

18 years old and above, 80 years old and below,

* Treated in the 3rd level intensive care unit for at least 48 hours,
* Not diagnosed with a psychiatric disease,
* Hemodynamically stable,
* Needing endotracheal aspiration,
* Not exposed to a painful procedure for at least one hour before the endotracheal aspiration procedure,
* Patients who do not receive high-dose inotropic support (Dopamine and/or Dobutamine 10 mcg/kg/hour) Patients who do not receive medical treatment for chronic pain
* Intubated and therefore unable to speak or verbally report pain, Ramsey Sedation Patients with 2 and 3 levels of alertness according to the scale

Exclusion Criteria:

Hearing problem,

* Having any limb, vascular problem or wound that prevents foot massage,
* Thrombophlebitis, occlusive artery disease, fever etc. It is inconvenient to apply massage due to illness,
* Endotracheal aspiration procedure (mouth/jaw/face etc. trauma, intracranial pressure being affected) is not applicable,
* Patients who did not agree to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Facial Anxiety Scale. | 30 minutes before tracheal aspiration; during tracheal aspiration;30 minutes after tracheal aspiration
  Facial Anxiety Scale was developed by Mckinley et al. (2003) to determine anxiety levels in intensive care patients. The scale consists of five different face types in the form of a card measuring 11x42 cm. While the anxiety level increases towards the face type in the left corner of the card, the anxiety level decreases towards the right corner. Anxiety face scale score evaluation is expressed as three points as medium level, three points above as high level, that is, three points and above as medium to high level.
Temperature will be measured from vital signs | 30 minutes before tracheal aspiration; during tracheal aspiration; 30 minutes after tracheal aspiration
  Body temperature will be measured with a thermometer device.
Measurement of the patient's pulse rate | 30 minutes before tracheal aspiration; during tracheal aspiration; 30 minutes after tracheal aspiration
  Pulse measurement will be measured with the help of a monitor.
Determination of respiratory rate | 30 minutes before tracheal aspiration; during tracheal aspiration; 30 minutes after tracheal aspiration
  The patient's respiratory rate will be measured with the help of a monitor.
Determination of the patient's blood pressure | 30 minutes before tracheal aspiration; during tracheal aspiration; 30 minutes after tracheal aspiration
  The patient's blood pressure will be measured with the help of a monitor.
Behavioral Pain Scale | 30 minutes before tracheal aspiration; during tracheal aspiration; 30 minutes after tracheal aspiration
  Behavioral Pain Scale (DAS) consists of three subscales, including facial expression,

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Tekinsoy Kartın, Ph.D, Principal Investigator — TC Erciyes University
Locations (2):
- Turkey (Türkiye) (2):
  - Pinar Tekinsoy Kartin, Melikgazi, Kayseri
  - Erciyes University, Kayseri, Melikgazi

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-11-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT06078826/SAP_000.pdf